CLINICAL TRIAL: NCT05981027
Title: Acute Effects of Static Stretching Exercises and the Mulligan Bent Leg Raise Technique on Hamstring Muscle Stiffness: an Ultrasound Elastography Evaluation
Brief Title: Static Stretching Exercises and Ultrasound Elastography Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Tahir Keskin , Pt, MSc, Research Assistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SuleymanDUtahirkeskin03
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Hamstring Muscle; Muscle Stretching Exercise; Elastography
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mulligan bent leg raise technique (Experimental): A single session of 3 repetitions of Mulligan bent leg raise was applied to the participants.
  Interventions: Other: Mulligan bent leg raise technique
- Static stretching exercise (Experimental): A single session of 5 repetitive stretching exercises was performed on the participants.
  Interventions: Other: Static stretching exercise

INTERVENTIONS:
Other: Mulligan bent leg raise technique — In this study, while the participant was lying on his back on a high bed, the physiotherapist sat on the lateral side of the leg to be treated, placing the popliteal fossa of the participant's knee on his shoulder. The hip and knee of the leg to be stretched were placed in 90° flexion. Distraction was applied to the lower end of the femur, and the participant was asked to push the physiotherapist's shoulder with his leg and then relax. At this relaxation point, the physiotherapist pushed the flexed knee as far as possible in the direction of the ipsilateral shoulder in a painless range.
  Arms: Mulligan bent leg raise technique
Other: Static stretching exercise — The participant lay on a stretcher in the supine position with his back straight. The physiotherapist placed the participant's leg on his shoulder with the knee in full extension and supported by the ankle and flexed the hip as much as possible until a tension was felt in the posterior thigh. This position was maintained for 30 seconds.
  Arms: Static stretching exercise

SUMMARY:
The aim of thid study was to compare two methods applied to increase the flexibility of the hamstring muscles and objectively evaluate changes in muscle stiffness using the two-dimensional shear wave ultrasound elastography (2D SWE) method. Thirty asymptomatic young individuals with hamstring shortness were divided into two groups by simple randomization. The Mulligan bent leg raise (BLR) technique was applied to the first group, and passive static stretching exercises to the second group. Hamstring flexibility was evaluated with the sit-and-reach test, and muscle stiffness with the 2D SWE method.

ELIGIBILITY:
Inclusion Criteria:

* Having a limitation of more than 25° in the active knee extension test
* Only engaged in recreational sports during the study period

Inclusion Criteria:

* Having a history of lower extremity injury within the last two years
* Not volunteering to participate in the study.

Ages: 20 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Back-saver sit-and-reach test | Up to 2 months
  The difference between the back-saver sit-and-reach test and the classical sit-and-reach test is that the former is applied unilaterally. The test was administered using the sit-and-reach test box. The participants were asked to sit on a flat surface and rest the sole of one of their feet flat on the end of the box while keeping the other leg flat on the floor by flexing the knee and hips to 90° and 45° sequentially. Maintaining this position, they were asked to place one hand on the other with their palms facing down, slide their hands on the measuring board, slowly reach forward, wait for a second or two at the last point reached

SECONDARY OUTCOMES:
Two-dimensional Shear Wave Elastography | Up to 2 months
  All 2D SWE examinations were performed by a specialist radiologist using the Philips EPIQ-7 (EPIQ Elite Diagnostic Ultrasound System Release 7.0.5 Philips) device with an 18-4 MHz linear probe. These measurements were made with the patient lying in the prone position, with the knees in full extension, the ankle at the end of the stretcher, and the feet hanging down. The probe was placed longitudinally in the middle 1/3 of the hamstring muscles. The participants were asked to keep their muscles in a relaxed position, and no extra pressure was applied to the probe to avoid tissue compression that could artificially affect the measured tissue stiffness

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No